CLINICAL TRIAL: NCT03259074
Title: A Randomized, Partially-blinded Study of Secukinumab to Demonstrate Reduction of Radiographic Progression Versus GP2017 (Adalimumab Biosimilar) at 104 Weeks and to Assess the Long Term Safety, Tolerability and Efficacy up to 2 Years in Patients With Active Ankylosing Spondylitis
Brief Title: Effect of Secukinumab on Radiographic Progression in Ankylosing Spondylitis as Compared to GP2017 (Adalimumab Biosimilar)
Acronym: SURPASS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAIN457K2340
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Results first posted 2023-03-09 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; AS; secukinumab; GP2017; adalimumab biosimilar; mSASSS; ASAS20; ASAS40; adult; r-axSpA; AIN457; radiographic; SURPASS
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — GP2017; adalimumab biosimilar HS016; secukinumab

STUDY DESIGN:
Intervention Model Description: Study was partially blinded. Subjects, investigators, site personnel, persons performing the assessments, monitors and the Sponsor remained blinded to the dose group of secukinumab (150 mg versus 300 mg)
Who Masked: Outcomes Assessor
Masking Description: The Participant, Care Provider, Investigator and Sponsor are blinded to Secukinumab dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AIN457 150 mg/placebo (Experimental): AIN457 150 mg and a matching placebo was administered subcutaneously via pre-filled syringes at Baseline, Weeks 1, 2, 3 and 4, followed by dosing every 4 weeks until Week 100
  Interventions: Biological: Placebo; Biological: AIN457 150 mg
- AIN457 300 mg (Experimental): AIN457 300 mg (2 x 150 mg) was administered subcutaneously via pre-filled syringes at Baseline, Weeks 1, 2, 3 and 4, followed by dosing every 4 weeks until Week 100
  Interventions: Biological: AIN457 150 mg
- GP2017 40mg (Active Comparator): GP2017 (adalimumab biosimilar) 40 mg was administered subcutaneously via pre-filled syringes at Baseline followed by dosing every 2 weeks until Week 102
  Interventions: Biological: GP2017 (adalimumab biosimilar)

INTERVENTIONS:
Biological: Placebo — Matching placebo to AIN457 150 mg dose administered with AIN457 via pre-filled syringes
  Arms: AIN457 150 mg/placebo
Biological: GP2017 (adalimumab biosimilar) — 40 mg in pre-filled syringes was administered subcutaneously
  Other Names: adalimumab biosimilar
  Arms: GP2017 40mg
Biological: AIN457 150 mg — 150 mg in pre-filled syringes was administered subcutaneously
  Other Names: secukinumab
  Arms: AIN457 150 mg/placebo; AIN457 300 mg

SUMMARY:
The purpose of this study is to demonstrate the impact of secukinumab on the progression of structural damage in the spine, as measured by the modified Stoke Ankylosing Spondylitis Spine Score (mSASSS) in patients with Ankylosing Spondylitis (AS).

DETAILED DESCRIPTION:
This was a Phase IIIb, multi-center, randomized, partially-blinded, active-controlled, parallel-group design in subjects with AS. The study consisted of a screening period (up to 10 weeks before randomization), a treatment period (104 weeks), and two follow-up visits (Weeks 112 and 120).

Subjects in both secukinumab dose groups received study treatment at baseline, Weeks 1, 2, 3 and 4 followed by treatment every 4 weeks through Week 100. Subjects in the GP2017 group received study treatment at baseline and every two weeks through Week 102. Subjects could self-administer all secukinumab / placebo and GP2017 doses at the study site or at home. Study treatment (secukinumab vs. GP2017) was provided in an open-label fashion. Subjects in the secukinumab groups were blinded to the dose (150 mg vs. 300 mg). Subjects who received rescue treatment with prohibited medications were allowed to remain in the study but had to discontinue study treatment. Subjects were treated for 104 weeks with two follow-up visits (Weeks 112 and 120).

A total of 859 subjects were randomized to treatment at 171 sites in 30 countries in Europe, North America, South America, and Asia.

.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-nursing female patients at least 18 years of age
* Diagnosis of moderate to severe Ankylosing Spondylitis with radiologic evidence (centrally read X-ray) fulfilling the Modified New York criteria for AS despite previous or current NSAID/ nonbiologic DMARD therapy
* Active AS assessed by total BASDAI ≥ 4 on a scale of 0-10
* Spinal pain as measured by BASDAI question #2 ≥ 4 (0-10)
* Total back pain as measured by visual analog scale (VAS) ≥ 40 mm (0-100 mm)
* hsCRP ≥ 5 mg/L OR presence of at least 1 syndesmophyte on centrally read spinal X-ray

Exclusion Criteria:

* Patients with total ankylosis of the spine
* Pregnant or nursing (lactating) women
* Evidence of ongoing infectious or malignant process
* Previous exposure to any biologic immunomodulating agent, including those targeting IL-17, IL-17 receptor or TNFα
* Subjects taking high potency opioid analgesics
* Previous treatment with any cell-depleting therapies including but not limited to anti-CD20, investigational agents

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 859 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (150):
- United States (19):
  - Novartis Investigative Site, Mesa, Arizona
  - Novartis Investigative Site, Escondido, California
  - Novartis Investigative Site, La Mesa, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Boise, Idaho
  - Novartis Investigative Site, Shreveport, Louisiana
  - Novartis Investigative Site, Wheaton, Maryland
  - Novartis Investigative Site, Great Falls, Montana
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Dayton, Ohio
  - Novartis Investigative Site, Middleburg Heights, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Mesquite, Texas
  - Novartis Investigative Site, Kennewick, Washington
  - Novartis Investigative Site, Franklin, Wisconsin
- Novartis Investigative Site, Ciudad Autonoma de Bs As, Argentina
- Novartis Investigative Site, Malvern East, Victoria, Australia
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Genk
- Canada (4):
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Barrie, Ontario
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Chile (3):
  - Novartis Investigative Site, Santiago, RM
  - Novartis Investigative Site, Concepción
  - Novartis Investigative Site, Santiago
- Colombia (2):
  - Novartis Investigative Site, Bucaramanga, Santander Department
  - Novartis Investigative Site, Barranquilla
- Czechia (4):
  - Novartis Investigative Site, Brno-Zidonice, CZE
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
- Denmark (2):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Copenhagen
- Novartis Investigative Site, Joensuu, Finland
- France (6):
  - Novartis Investigative Site, Nice, Cedex1
  - Novartis Investigative Site, Boulogne-Billancourt
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Monaco
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Germany (11):
  - Novartis Investigative Site, Bad Doberan
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Planegg
  - Novartis Investigative Site, Ratingen
- Greece (2):
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
- Israel (2):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Tel Aviv
- Japan (8):
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Nankoku, Kochi
  - Novartis Investigative Site, Tenri, Nara
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Meguro City, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
- Mexico (5):
  - Novartis Investigative Site, Torreón, Coahulia
  - Novartis Investigative Site, Mexicali, Estado de Baja California
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Culiacan, State of Mexico
  - Novartis Investigative Site, San Luis Potosí City
- Netherlands (5):
  - Novartis Investigative Site, Leiden, South Holland
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Leeuwarden
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Rotterdam
- Peru (4):
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, Santiago de Surco, Lima region
  - Novartis Investigative Site, Lima
- Philippines (2):
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Quezon City
- Poland (5):
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Dopiewo
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Sopot
- Portugal (5):
  - Novartis Investigative Site, Almada
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Ponte de Lima
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Vila Nova de Gaia
- Romania (2):
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
- Russia (11):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Ivanovo
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Slovakia (5):
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Piešťany, SVK
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Stará Ľubovňa
- South Korea (3):
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul
- Spain (12):
  - Novartis Investigative Site, Villajoyosa, Alicante
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, San Vicente de Barakaldo, Bizkaia
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, Vitoria-Gasteiz, Vitoria Gasteiz
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Taiwan (4):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Dalin
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Eskişehir
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli
- United Kingdom (14):
  - Novartis Investigative Site, Christchurch, Dorset
  - Novartis Investigative Site, London, Edmonton
  - Novartis Investigative Site, London, GBR
  - Novartis Investigative Site, Portsmouth, Hants
  - Novartis Investigative Site, Leytonstone, London
  - Novartis Investigative Site, Stoke-on-Trent, Staffordshire
  - Novartis Investigative Site, Bath
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Torquay
  - Novartis Investigative Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Sieper J, Poddubnyy D. Twenty years of clinical trials in axial spondyloarthritis: what can we learn for the future? Curr Opin Rheumatol. 2021 Jul 1;33(4):363-369. doi: 10.1097/BOR.0000000000000804. PMID 33978600
- [Derived] Baraliakos X, Ostergaard M, Gensler LS, Poddubnyy D, Lee EY, Kiltz U, Martin R, Sawata H, Readie A, Porter B; SURPASS Study Group. Comparison of the Effects of Secukinumab and Adalimumab Biosimilar on Radiographic Progression in Patients with Ankylosing Spondylitis: Design of a Randomized, Phase IIIb Study (SURPASS). Clin Drug Investig. 2020 Mar;40(3):269-278. doi: 10.1007/s40261-020-00886-7. PMID 31983056
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1307

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 859 subjects were randomized to treatment at 171 sites in 30 countries in Europe, North America, South America, and Asia
Groups:
- AIN457 150 mg/Placebo: AIN457 150 mg and a matching placebo was administered subcutaneously via pre-filled syringes at Baseline, Weeks 1, 2, 3 and 4, followed by dosing every 4 weeks until Week 104
- AIN457 300 mg: AIN457 300 mg (2 x 150 mg) was administered subcutaneously via pre-filled syringes at Baseline, Weeks 1, 2, 3 and 4, followed by dosing every 4 weeks until Week 104
- GP2017 40mg: GP2017 (adalimumab biosimilar) 40 mg was administered subcutaneously via pre-filled syringes at Baseline followed by dosing every 2 weeks until Week 104
Period: Overall Study
Arm/Group | AIN457 150 mg/Placebo | AIN457 300 mg | GP2017 40mg
Started | 287 | 286 | 286
Completed | 254 | 237 | 243
Not Completed | 33 | 49 | 43
Not completed — Adverse Event | 9 | 12 | 8
Not completed — Death | 1 | 1 | 3
Not completed — Lost to Follow-up | 2 | 4 | 3
Not completed — New Therapy For Study Indication | 1 | 2 | 2
Not completed — Physician Decision | 4 | 12 | 10
Not completed — Pregnancy | 1 | 1 | 0
Not completed — Progressive Disease | 1 | 0 | 0
Not completed — Protocol Deviation | 1 | 1 | 3
Not completed — Subject/Guardian Decision | 13 | 16 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 150 mg/Placebo | AIN457 300 mg | GP2017 40mg | Total
Number analyzed (Participants) | 287 | 286 | 286 | 859
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (11.99) | 42.2 (12.47) | 41.9 (12.68) | 42.1 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 63 | 65 | 185
  Male | 230 | 223 | 221 | 674
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 225 | 227 | 228 | 680
  Black or African American | 1 | 2 | 0 | 3
  Asian | 40 | 39 | 50 | 129
  American Indian or Alaska Native | 19 | 15 | 7 | 41
  Other | 1 | 0 | 0 | 1
  Multiple | 1 | 3 | 1 | 5
Modified Stoke Ankylosing Spondylitis Spine Score (mSASSS) scores [Mean (Standard Deviation); unit: score on a scale] — The modified Stoke Ankylosing Spondylitis Spine Score (mSASSS) evaluates the outside corners of the vertebral spine for erosions, sclerosis, squaring, bony growths and spinal bridging. The mSASSS assesses the participant's spinal vertebrae for structural changes and scores each vertebrae from 0 (normal vertebrae) to 3 (bony growth that bridges one vertebrae to the neighboring vertebrae). A total of 24 vertebral corners are scored for a possible maximum grade of 72. Population: The baseline mSASSS was determined only from those participants who provided evaluable baseline X-ray images.
  score on a scale
    number analyzed (Participants) | 283 | 280 | 283 | 846
    (all) | 17.602 (21.3286) | 16.527 (20.8153) | 15.695 (19.4955) | 16.609 (20.5506)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With no Radiographic Progression at Week 104 (Multiple Imputation) (Full Analysis Set)
Description: Radiographic progression was based on scores from the modified Stoke Ankylosing Spondylitis Spine Score (mSASSS). The mSASSS is the sum of scores assessing the vertebral corners of the lumbar and cervical spine as 0 (normal), 1 (erosion, sclerosis, or squaring), 2 (syndesmophyte), or 3 (bridging syndesmophyte) with a total range from 0-72. No radiographic progression was defined as the change from baseline in mSASSS score <= 0.5.
Time Frame: Baseline and at Week 104
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg/Placebo | AIN457 300 mg | GP2017 40mg
Number analyzed (Participants) | 287 | 286 | 286
Percentage of participants | 66.1 | 66.9 | 65.6
Statistical Analysis 1: Comparison: AIN457 150 mg/Placebo vs GP2017 40mg; Test type: Superiority; p = 0.7164, Regression, Logistic — Logistic regression model with treatment as a factor and baseline mSASSS score as a covariate using marginal standardization method; Marginal difference = 1.51, 95% CI 2-sided [-6.63 to 9.64]
Statistical Analysis 2: Comparison: AIN457 300 mg vs GP2017 40mg; Test type: Superiority; p = 0.6925, Regression, Logistic; Logistic regression model with treatment as a factor and baseline mSASSS score as a covariate using marginal standardization method; Marginal difference = 1.67, 95% CI 2-sided [-6.61 to 9.95]

2. Secondary Outcome: Change From Baseline in mSASSS at Week 104 (Multiple Imputation) (Full Analysis Set)
Description: Radiographic changes in the spine were based on the change in score of the modified Stoke Ankylosing Spondylitis Spinal Score (mSASSS) from baseline to Week 104.
  The mSASSS is the sum of scores assessing the vertebral corners of the lumbar and cervical spine as 0 (normal), 1 (erosion, sclerosis, or squaring), 2 (syndesmophyte), or 3 (bridging syndesmophyte) with a total range from 0-72.
Time Frame: Baseline and at Week 104
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mSASSS scores
Arm/Group | AIN457 150 mg/Placebo | AIN457 300 mg | GP2017 40mg
Number analyzed (Participants) | 287 | 286 | 286
mSASSS scores | 0.54 (0.175) | 0.55 (0.180) | 0.72 (0.177)
Statistical Analysis 1: Comparison: AIN457 150 mg/Placebo vs GP2017 40mg; Test type: Superiority — Due to to the pre-defined hierarchical testing strategy, p values beyond the primary endpoint which was not met were not presented; LS mean difference = -0.18, 95% CI 2-sided [-0.646 to 0.293] — ANCOVA model with treatment as a factor and baseline mSASSS score as a covariate
Statistical Analysis 2: Comparison: AIN457 300 mg vs GP2017 40mg; Test type: Superiority — [test comment as in outcome 2, analysis 1]; LS mean difference = -0.16, 95% CI 2-sided [-0.639 to 0.315] — ANCOVA model with treatment as a factor and baseline mSASSS score as a covariate

3. Secondary Outcome: Percentage of Participants Without New Syndesmophytes by mSASSS Between Baseline and Week 104 (Multiple Imputation) (Syndesmophyte Subset)
Description: Syndesmophytes are bony growths that develop on corner of the vertebrae of the spine which are indicators of AS. A participant was considered to have a syndesmophyte if at least one reader assessed vertebral corner as >= 2 at on the mSASSS scale at baseline. Only participants with a syndesmophyte at baseline were evaluated at Week 104 for new syndesmophytes. A new syndesmophyte was a syndesmophyte present at Week 104 which was not present at baseline. Absence of new syndesmophyte was defined as having individual vertebral score < 2 on the mSASSS scale for all interpretable locations that had no syndesmophyte at baseline. Missing responses for subjects without new syndesmophyte at Week 104 were imputed by multiple imputation (MCMC).
Time Frame: Baseline and at Week 104
Population: Syndesmophyte subset only included participants who had a syndesmophyte at baseline as measured on the mSASSS scale.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg/Placebo | AIN457 300 mg | GP2017 40mg
Number analyzed (Participants) | 211 | 204 | 212
Percentage of participants | 56.9 | 53.8 | 53.3
Statistical Analysis 1: Comparison: AIN457 150 mg/Placebo vs AIN457 300 mg; Test type: Superiority — [test comment as in outcome 2, analysis 1]; Marginal difference = 4.32, 95% CI 2-sided [-5.62 to 14.27] — Logistic regression model with treatment as a factor and baseline count of vertebral corners with syndesmophyte as a covariate using marginal standardization method
Statistical Analysis 2: Comparison: AIN457 300 mg vs GP2017 40mg; Test type: Superiority — [test comment as in outcome 2, analysis 1]; Marginal difference = 1.09, 95% CI 2-sided [-9.13 to 11.31] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline in MRI Berlin Sacroiliac (SI) Joint Edema Score (Observed Data) (MRI Subset)
Description: Magnetic Resonance Images (MRI) of the Sacroiliac Joint (SIJ) were assessed for the presence and severity of SIJ bone marrow edema according to the Berlin Active Inflammatory Lesions Scoring with a minimum score of 0 and a maximum score of 24. Higher scores indicate more inflammation.
Time Frame: Baseline and at Week 104
Population: MRI subset only included participants who had an MRI performed at selected centers
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 150 mg/Placebo | AIN457 300 mg | GP2017 40mg
Number analyzed (Participants) | 137 | 137 | 144
scores on a scale | -1.527 (0.1057) | -1.378 (0.1097) | -1.710 (0.1087)
Statistical Analysis 1: Comparison: AIN457 150 mg/Placebo vs GP2017 40mg; Week 104 - 150 mg; Test type: Other — [test comment as in outcome 2, analysis 1]; LS Means = 0.183, 95% CI 2-sided [-0.12 to 0.48], Standard Error of Mean 0.1517 — LS Means and 95% CI are from an ANCOVA model with treatment as a factor, baseline Berlin SI joint edema score as a covariate
Statistical Analysis 2: Comparison: AIN457 300 mg vs GP2017 40mg; Week 104 - 300 mg; Test type: Other — [test comment as in outcome 2, analysis 1]; LS Means = 0.332, 95% CI 2-sided [0.03 to 0.64], Standard Error of Mean 0.1545 — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline in Berlin Modification of ASspiMRI-a Edema Score (MRI Subset)
Description: Magnetic Resonance Images (MRI) of the spine were assessed for the presence and severity of bone marrow edema in the spinal vertebrae according to the Berlin modification of the ASspiMRI-a edema score with a score range of 0 to 69. Higher scores indicate more inflammation.
Time Frame: Baseline and at Week 104
Population: MRI subset only included participants who had an MRI performed at selected centers
Measure: Least Squares Mean (Standard Error); unit: Berlin mod. of ASspiMRI-a edema scores
Arm/Group | AIN457 150 mg/Placebo | AIN457 300 mg | GP2017 40mg
Number analyzed (Participants) | 137 | 137 | 144
Berlin mod. of ASspiMRI-a edema scores | -1.224 (0.2306) | -1.683 (0.2373) | -2.101 (0.2378)
Statistical Analysis 1: Comparison: AIN457 150 mg/Placebo vs GP2017 40mg; Week 104 - 150 mg; Test type: Other — [test comment as in outcome 2, analysis 1]; LS Means = 0.877, 95% CI 2-sided [0.22 to 1.53], Standard Error of Mean 0.3316 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: AIN457 300 mg vs GP2017 40mg; Week 104 - 300 mg; Test type: Other — [test comment as in outcome 2, analysis 1]; LS Means = 0.419, 95% CI 2-sided [-0.24 to 1.08], Standard Error of Mean 0.3357 — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Percentage of Responders for Assessment of SpondyloArthritis International Society 20 (ASAS20)
Description: Assessment of SpondyloArthritis International Society criteria (ASAS) consist of 4 domains measured on visual analog scales (VAS): 1. Patient's global assessment; 2. Patient's assessment of back pain; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). ASAS 20 response is defined as an improvement of ≥20% and ≥1 unit on a scale of 10 in at least three of the four main domains and no worsening of ≥20% and ≥1 unit on a scale of 10 in the remaining domain. A higher score on the VAS signifies higher severity.
Time Frame: Week 104
Population: Full analysis set for the population to be analyzed in this secondary outcome: AIN457 150 mg and AIN457 300 mg arms.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AIN457 150 mg/Placebo | AIN457 300 mg
Number analyzed (Participants) | 287 | 286
Percentage of participants | 83.1 [77.8 to 87.4] | 82.9 [77.3 to 87.4]
Statistical Analysis 1: Comparison: AIN457 150 mg/Placebo vs AIN457 300 mg; Test type: Other — [test comment as in outcome 2, analysis 1]; Marginal difference = 1.54, 95% CI 2-sided [-5.10 to 8.18] — Estimated mean, marginal difference and 95% confidence interval are from a logistic regression model with treatment as a factor using marginal standardization method

7. Secondary Outcome: Percentage of Responders for Assessment of SpondyloArthritis International Society 40 (ASAS 40)
Description: Assessment of SpondyloArthritis International Society criteria (ASAS) consist of 4 domains measured on visual analog scales (VAS): 1. Patient's global assessment; 2. Patient's assessment of back pain; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). ASAS40 response is defined as an improvement of ≥40% and ≥2 units on a scale of 10 in at least three of the four ASAS main domains and no worsening at all in the remaining domain. A higher score on the VAS signifies higher severity.
Time Frame: Week 104
Population: Full analysis set for the population to be analyzed in this secondary outcome: AIN457 150 mg and AIN457 300 mg arms.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AIN457 150 mg/Placebo | AIN457 300 mg
Number analyzed (Participants) | 287 | 286
Percentage of participants | 69.9 [63.7 to 75.4] | 73.5 [67.3 to 78.9]
Statistical Analysis 1: Comparison: AIN457 150 mg/Placebo vs AIN457 300 mg; Test type: Other — [test comment as in outcome 2, analysis 1]; Marginal difference = -2.34, 95% CI 2-sided [-10.18 to 5.51] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Percentage of Responders for Assessment of SpondyloArthritis International Society With a Partial Remission Response (Full Analysis Set)
Description: The Assessment of SpondyloArthritis International Society (ASAS) partial remission response criteria consisted of the following assessment domains measured on visual analogue scales (VAS): 1. Patient's global assessment; 2. Patient's assessment of back pain; 3. Function represented by BASFI average of 10 questions regarding ability to perform specific tasks; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). The ASAS partial remission criteria was defined as a value not above 2 units in each of the four domains on a scale of 10.
Time Frame: Week 104
Population: Full analysis set for the population to be analyzed in this secondary outcome: AIN457 150 mg and AIN457 300 mg arms.
Measure: Number (95% Confidence Interval); unit: Percentage participants
Arm/Group | AIN457 150 mg/Placebo | AIN457 300 mg
Number analyzed (Participants) | 287 | 286
Percentage participants | 31.5 [25.9 to 37.7] | 30.2 [24.5 to 36.6]
Statistical Analysis 1: Comparison: AIN457 150 mg/Placebo vs AIN457 300 mg; Test type: Other — [test comment as in outcome 2, analysis 1]; Marginal difference; Marginal difference = 2.18, 95% CI 2-sided [-5.34 to 9.69] — [estimate comment as in outcome 6, analysis 1]

9. Secondary Outcome: Percentage of Participants With Assessment of SpondyloArthritis International Society for Inactive Disease Response (Observed Data) (Full Analysis Set)
Description: The Ankylosing Spondylitis Disease Activity Score (ASDAS) is a composite index to assess disease activity in AS. Parameters used for the ASDAS include spinal pain (BASDAI question 2), the patient's global assessment of disease activity, peripheral pain/swelling (BASDAI question 3), duration of morning stiffness (BASDAI question 6) and C-reactive protein (CRP) in mg/L (Sieper 2009, Lukas 2009). Disease activity states are inactive disease, moderate disease activity, high disease activity, and very high disease activity. The 3 values selected to separate these states were < 1.3 between inactive disease and moderate disease activity, < 2.1 between moderate disease activity and high disease activity, and > 3.5 between high disease activity and very high disease activity. Selected cutoffs for improvement scores were a change ≥ 1.1 unit for "minimal clinically important improvement" and a change ≥ 2.0 units for "major improvement" (Machado 2011).
Time Frame: Week 104
Population: Full analysis set for the population to be analyzed in this secondary outcome: AIN457 150 mg and AIN457 300 mg arms.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AIN457 150 mg/Placebo | AIN457 300 mg
Number analyzed (Participants) | 287 | 286
Percentage of participants | 31.1 [25.5 to 37.4] | 31.7 [25.7 to 38.3]
Statistical Analysis 1: Comparison: AIN457 150 mg/Placebo vs AIN457 300 mg; Test type: Other; Due to to the pre-defined hierarchical testing strategy, p values beyond the primary endpoint which was not met were not presented; Marginal difference = 0.33, 95% CI 2-sided [-7.08 to 7.74] — [estimate comment as in outcome 6, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 84 days up to a maximum of 900 days for AIN 457 and 939 days for GP2017.
Groups:
- GP2017 40 mg: GP2017 (adalimumab biosimilar) 40 mg was administered subcutaneously via pre-filled syringes at Baseline followed by dosing every 2 weeks until Week 104
Arm/Group | AIN457 150 mg/Placebo | AIN457 300 mg | GP2017 40 mg
All-Cause Mortality (participants affected / at risk) | 1/286 | 1/285 | 3/285
Serious Adverse Events (participants affected / at risk) | 40/286 | 29/285 | 32/285
Other Adverse Events (participants affected / at risk) | 106/286 | 107/285 | 99/285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 150 mg/Placebo (N=286) | AIN457 300 mg (N=285) | GP2017 40 mg (N=285)
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Iridocyclitis (Eye disorders) | 2 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 3 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 2 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Ileal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 2
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 1 | 0
Drug intolerance (General disorders) | 1 | 0 | 0
Medical device pain (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Immunosuppression (Immune system disorders) | 0 | 1 | 0
Abscess intestinal (Infections and infestations) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Myelitis (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 2
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain hypoxia (Nervous system disorders) | 0 | 0 | 1
Facial paresis (Nervous system disorders) | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 1
Lacunar stroke (Nervous system disorders) | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 1
Device issue (Product Issues) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1
Depression suicidal (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 1
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 1 | 0
Iliac artery stenosis (Vascular disorders) | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 150 mg/Placebo (N=286) | AIN457 300 mg (N=285) | GP2017 40 mg (N=285)
Diarrhoea (Gastrointestinal disorders) | 20 | 22 | 11
Nasopharyngitis (Infections and infestations) | 47 | 40 | 44
Upper respiratory tract infection (Infections and infestations) | 17 | 25 | 18
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 11 | 17 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 13 | 12
Headache (Nervous system disorders) | 16 | 17 | 17
Hypertension (Vascular disorders) | 11 | 11 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT03259074/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT03259074/SAP_001.pdf